CLINICAL TRIAL: NCT06088563
Title: Study of the Impact of Time of Vaccination on Response to Influenza Vaccine in Kidney Transplant Recipients -ChronoVAX
Acronym: CHRONOVAX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23-PP-09
Record Dates: First submitted 2023-10-06; First posted 2023-10-18 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Vaccination; Infection
Keywords: Influenza; Kidney transplant; Vaccination
MeSH Terms: conditions — Infections; Influenza, Human | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning injection (Active Comparator): EFLUELDA influenza vaccine injection between 07:00 am and 09:00 am.
  Interventions: Other: Vaccine injection
- Evening injection (Active Comparator): EFLUELDA influenza vaccine injection between 07:00 pm and 09:00 pm.
  Interventions: Other: Vaccine injection

INTERVENTIONS:
Other: Vaccine injection — Injection of the vaccine in renal transplant patients.
  Other Names: EFLUELDA - Fluzone High-Dose Quadrivalent

SUMMARY:
Immune response to influenza vaccine in kidney transplant patients

DETAILED DESCRIPTION:
Seasonal influenza vaccination is recommended for kidney transplant patients, as influenza is responsible for significant morbidity and mortality in this immunocompromised population. Nevertheless, injection of influenza vaccine induces a protective immune response in only 20% to 40% of patients. Today, there are no recommendations regarding the injection time of influenza vaccine in the general population or in immunocompromised patients. In this context, recent studies conducted in healthy subjects have shown that the time of vaccination can have an impact on vaccine efficacy. This is the case for BCG, influenza, COVID-19. On this basis, we formulate the main hypothesis that the administration of influenza vaccine to kidney transplant patients would be more effective when carried out in the morning than in the evening.

ELIGIBILITY:
Inclusion Criteria:

* Renal transplant patient;
* Follow-up at Nice University Hospital;
* Age > 18 years;
* Indication for influenza vaccination
* Free and informed consent;
* Immunosuppressive treatment including anti-calcineurin and/or Mycophenolate Mofetil (with or without corticoids).

Exclusion Criteria:

* Known hypersensitivity to influenza vaccine or egg proteins;
* Influenza vaccination for the 2023-2024 season already performed;
* Current infection;
* Current acute medical condition;
* Treatment of rejection within the previous 3 months;
* Immunosuppressive therapy including CTLA4 agonist, mTOR inhibitor, complement inhibitor, anti-CD19;
* Polyvalent immunoglobulin infusion within the preceding 3 months;
* Vulnerable persons (minors, adults under guardianship or trusteeship, pregnant women, persons deprived of their liberty, persons unable to speak French);
* Subjects not affiliated to the Social Security system.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-10-26 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Comparison of antibody titer (seroconversion) 4 weeks after inactivated influenza vaccine injection in each arm. | 7 months
  Seroconversion will be defined as an increase in antibody titer of at least 4-fold (≥4) over pre-vaccination titer AND an antibody titer ≥ 1:40 (seroprotection) four weeks post-vaccination, for at least one of the three vaccine antigens.

SECONDARY OUTCOMES:
Number of seasonal influenza virus infections in each arm. | 8 months
  Comparing the number of seasonal influenza virus infections in kidney transplant patients between a group of patients vaccinated in the morning and a group vaccinated in the evening.
  The occurrence of influenza, as confirmed by a PCR test, will be noted in the follow-up consultation.
Comparison the evolution of antibody titres reacting in each arm. | 7 months
  In kidney transplant patients, compare the evolution of antibody titres reacting with vaccine antigens 4 weeks after influenza vaccination between a group of patients vaccinated in the morning and a group of patients vaccinated in the evening.
  The titer of antibodies reacting with vaccine antigens is measured by ELISA ;
Evolution of the number of memory B cells in each arm. | 7 months
  To compare in kidney transplant patients the evolution of the number of memory B cells reacting with vaccine antigens 4 weeks after influenza vaccination between a group of patients vaccinated in the morning and a group of patients vaccinated in the evening.
  The number of memory B cells reacting with vaccine antigens will be measured by ELISPOT ;
Evolution of the number of CD4+ T cells in each arm. | 7 months
  Comparing the evolution of CD4+ T cells reacting with vaccine antigens in kidney transplant patients 4 weeks after influenza vaccination between a group of patients vaccinated in the morning and a group of patients vaccinated in the evening.
  The number of CD4+ T cells reacting with vaccine antigens will be measured by in vitro proliferation assay;
Evolution of the number of CD8+ T cells in each arm. | 7 months
  Comparing the evolution of CD8+ T cells reacting with vaccine antigens in kidney transplant patients 4 weeks after influenza vaccination between a group of patients vaccinated in the morning and a group of patients vaccinated in the evening.
  The number of CD8+ T cells reacting with vaccine antigens will be measured by in vitro proliferation assay;

CONTACTS AND LOCATIONS:
Overall Officials: GOSSET Clément, MD, Principal Investigator — CHU NICE
Locations (1):
- CHU Nice - Hôpital Pasteur 2, Nice, Alpes-Maritimes, France

IPD SHARING:
Plan to Share IPD: No